CLINICAL TRIAL: NCT06126848
Title: Early Detection of Health Deterioration in Elderly Patients After Hospitalization for Heart Failure Decompensation: A Potential Role for Ambient Sensor Systems in the Patients Home
Brief Title: Early Detection of Health Deterioration in Elderly Patients After Hospitalization for Heart Failure Decompensation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nisha Arenja (Other)
Responsible Party: Sponsor-Investigator, Nisha Arenja, Pinciple Investigator, Kantonsspital Olten
Organization: Kantonsspital Olten (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: eHealth-HF
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation Cohort (Other)
  Interventions: Device: Ambient sensor system

INTERVENTIONS:
Device: Ambient sensor system — Main study: A contactless non-intrusive ambient sensor system including infrared motion sensors combined with a contactless Emfit bed sensor will be installed in the home of single living study patients by using a commercially available System (Domo Health®, Lausanne) after informed consent has been obtained. Sensor data are prospectively followed over 3-6 months for predefined indicators of health deterioration. If indicators for health deterioration are present, patients will be called in to the hospital for cardiology consult by the study team including blood analysis for follow-up of BNP values and if necessary, therapy adaption.

SUMMARY:
Digital biomarkers extracted by ambient sensor signals are a promising tool for early detection of health deterioration in the setting of remote patient management of heart failure patients.The primary objective of the study is to evaluate new digital biomarkers as predictors of impending heart failure decompensation.

Secondary objectives are (1) outcome assessment (re-hospitalizations, cardiovascular death, all-cause death), (2) quality of life and (3) System User Satisfaction (SUS)

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital for worsening HF
* age ≥ 70 years
* LVEF < 50% and need of diuretics
* NYHA II or III
* living alone
* willing to participate with informed consent.

Exclusion Criteria:

* Major depression (PHQ 9-score >9)
* being on hemodialysis
* had been admitted to hospital for any reason within 7 days before HF decompensation.
* patients with a left ventricular assist device
* coronary revascularization or cardiac resynchronization therapy implantation within 28 days before the index event of HF decompensation or have been scheduled for such interventions.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of ambient sensor derived digital biomarkers | 6 months
  Sensitivity and specificity of a combination of ambient sensor derived digital biomarker for the prediction of brain natriuretic peptide (BNP) increase of ≥ 20% compared to baseline value.

SECONDARY OUTCOMES:
Outcome assessment | 6 months
  re-hospitalizations, cardiovascular death, all-cause death
Quality of life (heart failure symptoms) - KCCQ | 6 months
  KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
System Usability Scale (SUS) | 6 months
  SUS score 0-100; 80.3 or higher is an A. People will recommend it to their friends 68 or there abouts gets you a C. You are doing OK but could improve 51 or under gets you a big fat F. Make usability your priority now and fix this fast.

REFERENCES:
- [Derived] Haas K, Scheidegger-Balmer F, Meichtry A, Vogeli B, Arenja N, Buluschek P, Saner H. Association Between Refrigerator Openings and Protein Intake After Hospitalization for Heart Failure Decompensation: Protocol for a Prospective Cohort Pilot Study. JMIR Res Protoc. 2025 Aug 18;14:e66299. doi: 10.2196/66299. PMID 40824685
- [Derived] Vogeli B, Arenja N, Schutz N, Nef T, Buluschek P, Saner H. Evaluation of Ambient Sensor Systems for the Early Detection of Heart Failure Decompensation in Older Patients Living at Home Alone: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2024 May 31;13:e55953. doi: 10.2196/55953. PMID 38820577